CLINICAL TRIAL: NCT00352287
Title: Effects of GH and Pioglitazone in Viscerally Obese Adults With IGT
Brief Title: Study to Determine the Effects of Human Growth Hormone and Pioglitazone in Overweight, Prediabetic Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 78235; 1F32-AG02142-1, 5F32-AG02142-2
Record Dates: First submitted 2006-07-12; First posted 2006-07-14 (Estimated); Last update posted 2006-07-14 (Estimated); Status verified 2006-07

CONDITIONS: Obesity; Metabolic Syndrome; Impaired Glucose Tolerance
Keywords: Visceral fat; Impaired glucose tolerance; Insulin resistance; Growth hormone; Thiazolidinedione
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Glucose Intolerance; Insulin Resistance | interventions — Growth Hormone; Pioglitazone

INTERVENTIONS:
Drug: Recombinant human growth hormone; pioglitazone

SUMMARY:
The purpose of the study was to determine the effects of growth hormone and an insulin sensitizer drug in pre-diabetic adults with excessive amounts of abdominal fat. Participants received a combination of two drugs: (1) recombinant human growth hormone (or its placebo) and (2) pioglitazone (or its placebo). We measured the abdominal fat content and blood sugar levels of participants before and after 40 weeks of treatment.

DETAILED DESCRIPTION:
Treatment with recombinant human growth hormone (GH) has been shown to reduce visceral adipose tissue (VAT) and improve insulin sensitivity in normoglycemic adults, but glucose levels may rise transiently. Pioglitazone, a thiazolidinedione (TZD) drug, counters the short-term diabetogenic effect of GH in rodents, but combined use of these drugs has not been evaluated in humans.

The purpose of this study was to determine the effects of GH and a TZD, alone and in combination, on glucose metabolism, visceral adiposity and insulin sensitivity in abdominally obese adults with impaired glucose tolerance. The hypothesis that combined treatment attenuates GH-induced increases in glucose concentrations, reduces VAT, and improves insulin sensitivity over time was tested. Sixty-two adults received GH and pioglitazone for 40 weeks in a double-blind, randomized, placebo-controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 75 years
* BMI > 27 kg/m2
* Waist circumference >100 cm for men and > 88 cm for women
* Impaired glucose tolerance (documented by a 75 gram OGTT)

Exclusion Criteria:

* Diabetes mellitus
* Malignancy
* Premenopausal women who are breastfeeding or decline contraception
* Congestive heart failure
* ALT > 3 times upper normal limit

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-03; Study Completion 2005-04

PRIMARY OUTCOMES:
Visceral fat content was quantified by CT scan, glucose tolerance was assessed using a 75 gm OGTT and insulin sensitivity was measured using steady-state plasma glucose (SSPG) levels obtained during an insulin suppression test.

SECONDARY OUTCOMES:
Body mass index (BMI), anthropometric measurements, glycohemoglobin and lipid measurements were performed before and after 40 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R Hoffman, MD, Principal Investigator — Stanford University; Hamdee Y Attallah, MD, Principal Investigator — Wayne State University
Locations (1):
- Veterans Affairs Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Derived] Ipsen EO, Madsen KS, Chi Y, Pedersen-Bjergaard U, Richter B, Metzendorf MI, Hemmingsen B. Pioglitazone for prevention or delay of type 2 diabetes mellitus and its associated complications in people at risk for the development of type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 19;11(11):CD013516. doi: 10.1002/14651858.CD013516.pub2. PMID 33210751